The Use of Delta-Wave Hypnoanalgesia as a Non-Pharmacological Adjunct to Reduce Perioperative Anxiety During Cataract Surgery: A Prospective Randomized Single-Blind Study

## **Consent Form for Participation in Clinical Research**

| Title of the Study: Perioperative Auditory Hypnoanaigesia in Cataract Surgery. |
|---|
| I, the undersigned, hereby agree to participate in the study entitled: "Perioperative Auditory Hypnoanalgesia in Cataract Surgery." |
| The objectives and procedures of the study have been clearly explained to me by Doctors Haythem ElAskri and Eslem Berrima. |
| I have read and understood the information sheet that was provided to me. |
| I agree that the documents from my medical record related to the study may be accessed by<br>the study investigators and, if necessary, by health authorities. Apart from these individuals,<br>who will handle the information with the strictest confidentiality, my anonymity will be<br>preserved. |
| I fully understand that my participation in the study is voluntary. I am free to accept or refuse to participate, and this will not affect the quality of care I receive. |
| My consent does not absolve the organizers of this study from their responsibilities. I retain all rights protected by law. |
| After discussing the study and receiving answers to all my questions, I freely and voluntarily agree to participate in the proposed research. |
| Done atOn |
| Name and signature of the participan |